CLINICAL TRIAL: NCT05537064
Title: A Pilot Study of Strategies to Increase Use of Centralized Pharmacy Services for Management of Statin Therapy Among Patients With or at High Risk for Atherosclerotic Vascular Disease
Brief Title: Centralized Prescribing for Statins
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 851668
Record Dates: First submitted 2022-09-07; First posted 2022-09-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Control arm exposed only to usual care, which consists of the passive decision support functionality Health Maintenance flag that is the current decision-support tool in the EMR.
- Non-visit Based Intervention (Experimental): In this arm the investigators will evaluate a non-visit-based nudge to refer patients eligible for but not prescribed high-intensity statins to centralized pharmacy services for initiation and/or titration of a statin. Practices will be randomized to usual care versus the non-visit-based nudge. The non-visit-based nudge will consist of an EPIC In-basket message sent to each provider that identifies their patients eligible for but not prescribed high- or moderate-intensity statins and notifies them that pended orders for a referral to centralized pharmacy services for statin management will be entered for these patients unless the provider opts out. At the time the in-basket message is sent out, PCPs will also have the opportunity to opt out of participating in the trial entirely.
  Interventions: Behavioral: Non-visit Based Intervention
- Visit-Based Intervention (Experimental): In this arm the investigators will evaluate a visit-based nudge to refer to centralized pharmacy services to refer patients eligible for but not prescribed high-intensity statins to centralized pharmacy services for initiation and/or titration of a statin. Physicians in a single practice will be randomized to usual care versus visit-based nudge. The visit-based nudge will consist of an interruptive Best Practice Advisory (BPA) in the EMR that will trigger during non-acute patient visits and will prompt the provider to refer the patient to a centralized pharmacy service for statin initiation and management.
  Interventions: Behavioral: Visit-Based Intervention

INTERVENTIONS:
Behavioral: Non-visit Based Intervention — At the beginning of the study period, PCPs will be sent an Inbasket message, a secure electronic messaging system included in EPIC, similar to an email. The message will notify them that pended orders for a referral to centralized pharmacy services for statin management will be entered for eligible patients unless the provider opts out. If no opt-out is received from the PCP within 7 days of receiving the message, their eligible patient panels will be referred to a centralized pharmacy team to begin pending referral orders to the PCP for eligible patients. Pharmacists affiliated with the centralized pharmacy service will then enter pended orders for referral to centralized pharmacy services that PCPs can sign either individually or in bulk. After the PCP signs the order for referral to centralized pharmacy services, a pharmacist from the centralized pharmacy team will then reach out to the patient on behalf of their PCP and discuss their indication for statin therapy.
  Arms: Non-visit Based Intervention
Behavioral: Visit-Based Intervention — The study team will build an interruptive BestPractice advisory (BPA), a pop-up notification in the EHR that is delivered to the PCP when they open the patient's chart during a non-acute patient visit. The BestPractice Advisory will describe the guideline criteria for which the patient is eligible for statin therapy, and recommend referral to a centralized pharmacy service for statin initiation and management. It will also include a link to a menu for prescribing an appropriate-dose statin, should the PCP want to prescribe a statin without referral to pharmacy services. The option for ordering referral to centralized pharmacy services will be pre-selected, such that if the PCP simply clicks "Accept" on the BPA, an order for referral to centralized pharmacy services for statin initiation and management will be generated.
  Arms: Visit-Based Intervention

SUMMARY:
This pilot study consists of a pair of pragmatic clinical trials that will evaluate two separate methods for optimizing referral of eligible patients to a centralized pharmacy service for statin management: 1) A stepped wedge clinical trial, with randomization at the level of the provider, evaluating a visit-based nudge for referral to pharmacy services versus usual care; 2) A cluster randomized trial, with randomization at the level of the practice, evaluating a non-visit based nudge for referral to pharmacy services versus usual care.

DETAILED DESCRIPTION:
This pilot study consists of a pair of pragmatic clinical trials that will evaluate two separate methods for optimizing referral of eligible patients to a centralized pharmacy service for statin management: 1) A stepped wedge clinical trial, with randomization at the level of the provider, evaluating a visit-based nudge for referral to pharmacy services versus usual care; 2) A cluster randomized trial, with randomization at the level of the practice, evaluating a non-visit based nudge for referral to pharmacy services versus usual care.

For trial #1, the investigators will identify PCPs at a single practice with at least 10 patients on their panel who are eligible for but not yet prescribed high- or moderate-intensity statin medication. These physicians will be randomized in stepped-wedge fashion to usual care or to a nudge, delivered at the time of a scheduled office visit, to refer appropriate patients to centralized pharmacy services for initiation and/or titration of a statin medication. In trial #2, the investigators will identify PCPs at 12 practices with at least 10 patients on their panel who are eligible for but not yet prescribed high- or moderate-intensity statin medication. Practices will be randomized to usual care or to a non-visit-based nudge to refer appropriate patients to centralized pharmacy services for initiation and/or titration of a statin medication. It is estimated that 13 practices and 83 providers will be eligible to participate in the two trials. The invesitgators will run the intervention over a 9-month time frame.

The primary outcome is the prescription of a statin for eligible patients during the 9-month timeframe. Secondary outcomes will include the prescription of guideline-directed intensity of statin medications as well as statin pharmacy dispense rate. The investigators will also assess LDL control over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Providers with at least 10 patients among their entire panel who meet the following criteria:
* Have a LGH PCP, AND
* 21-75 years old, AND
* An indication for high- or moderate-intensity statin, AND

  * Pooled cohort risk equation 10-year ASCVD risk greater than 10%, OR
  * diabetes mellitus, OR
  * very high LDL-C > 190 mg/dL, OR
  * familial hyperlipidemia, OR
  * established ASCVD,
* Not currently on statin therapy, OR on low dose-statin therapy

Exclusion Criteria:

* Have an allergy to statins
* Severe renal insufficiency defined as glomerular filtration rate (GFR) less than 30 mL/min or on dialysis
* Adverse reaction to statins including statin-related a) myopathy; b) Rhabdomyolysis; c) hepatitis
* Pregnant
* Currently breastfeeding
* On hospice or at the end-of-life
* On a PCSK9 Inhibitor medication
* Physicians (and their respective patients) will be excluded if they have less than 10 patients among their entire panel that are eligible for a statin medication.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1950 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Prescribed a Statin (population level) | 9 months
  The primary outcome is the prescription of a statin for eligible patients during the 9-month timeframe, assessed among all patients assigned to the physician or office eligible for but not prescribed a high-intensity statin at the start of the trial. The primary outcome will be compared between patients seeing physicians, or seen at practices, randomized to the intervention vs. usual care.
Number of Participants Prescribed a Statin (office-visit level) | 9 months
  The primary outcome is the prescription of a statin for eligible patients during the 9-month timeframe, assessed among all patients who had an office visit during the study period and were eligible for but not prescribed a high-intensity statin at the start of the trial. The primary outcome will be compared between patients seeing physicians, or seen at practices, randomized to the intervention vs. usual care.

SECONDARY OUTCOMES:
Statin Pharmacy Dispense Rate | 9 months
  Secondary outcomes will include the prescription of guideline-directed intensity of statin medications as well as statin pharmacy dispense rate. We will compare the proportion of eligible patients prescribed a guideline-concordant-intensity statin and the proportion filling a prescription for statin between patients seeing physicians randomized to intervention vs. usual care. This analysis will be performed both on the population-level (all patients assigned to the practice or physician eligible for but not prescribed a high-intensity statin at the start of the trial) and among patients with an office visit during the study period.

OTHER OUTCOMES:
LDL Control | 9 months
  We will also assess LDL control over the study period. We will compare the LDL between patients seeing physicians randomized to intervention vs. usual care. This analysis will be performed both on the population-level (all patients assigned to the practice or physician eligible for but not prescribed a high-intensity statin at the start of the trial) and among patients with an office visit during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fanaroff, MD, MHS, Principal Investigator — University of Pennsylvania
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

REFERENCES:
- [Derived] Fanaroff AC, Huang Q, Clark K, Norton LA, Kellum WE, Eichelberger D, Wood JC, Bricker Z, Dooley Wood AG, Kemmer G, Smith JI, Adusumalli S, Putt ME, Volpp KG. Encouraging Pharmacist Referrals for Evidence-Based Statin Initiation: Two Cluster Randomized Clinical Trials. JAMA Cardiol. 2025 May 1;10(5):473-481. doi: 10.1001/jamacardio.2025.0244. PMID 40136263
- [Derived] Fanaroff AC, Huang Q, Clark K, Norton LA, Kellum WE, Eichelberger D, Wood JC, Bricker Z, Wood AGD, Kemmer G, Smith JI, Adusumalli S, Putt M, Volpp KGM. Two randomized controlled trials of nudges to encourage referrals to centralized pharmacy services for evidence-based statin initiation in high-risk patients: Rationale and design of the SUPER LIPID program. Am Heart J. 2024 Jul;273:83-89. doi: 10.1016/j.ahj.2024.04.013. Epub 2024 Apr 26. PMID 38679189